CLINICAL TRIAL: NCT07190573
Title: Head and Neck Cancer Omics-integrated Precision mEdicine (HOPE)
Brief Title: Head and Neck Cancer Omics/Integrated Precision Medicine (HOPE)
Acronym: HOPE
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Nayeon Choi, Coordinatr, Head and Neck Cancer Center; Assitant Professor, Department of Otorhinolaryngology, Samsung Medical Center/Sungkyunkwan University School of Medicine, Samsung Medical Center
Other Study IDs: 2025-02-141
Record Dates: First submitted 2025-09-03; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer; squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Tissue: Fresh tissue will be collected whenever feasible. Residual samples from diagnostic or therapeutic biopsies and surgical resections will also be utilized. Additional residual tissue may be obtained during follow-up biopsies performed for suspected recurrence or treatment response assessment. At the time of surgery, tumor tissue, adjacent normal tissue, distant normal tissue, and lymph nodes will be collected.
  Blood: Peripheral blood will be collected at defined timepoints: prior to treatment, during treatment (for CCRT: baseline, 3 ± 1 weeks, 6 ± 1 weeks; for immunotherapy: baseline, 3 ± 1 weeks, 6 ± 1 weeks, 12 ± 3 weeks), during follow-up imaging, and at disease progression. Each draw will obtain 20-30 mL.
  Storage: All tissue and blood specimens will be stored in a designated, secure cryogenic facility, strictly for research purposes, without compromising clinical diagnosis or treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study Background and Rationale Head and neck cancer (HNC) is the sixth leading cause of cancer-related death, with over 650,000 new cases diagnosed worldwide each year. About 60% of patients are diagnosed at an advanced stage, and many experience recurrence or spread despite surgery, radiation, or chemotherapy. Major risk factors include tobacco and alcohol use, prior radiation therapy, and infection with human papillomavirus (HPV).

The prognosis differs across patients due to HPV infection and genetic factors. HPV is commonly found in cancers of the tonsils and throat. Patients with HPV-positive tumors generally respond better to treatment and live longer than those who are HPV-negative. Conversely, patients with certain genetic changes, like EGFR amplification, tend to have worse outcomes.

HNC can develop in the oral cavity, throat, larynx, nasal cavity, nasopharynx, and salivary glands. Squamous cell carcinoma caused by smoking is the most common type, but other types like salivary gland cancer or adenoid cystic carcinoma also occur, making the disease clinically diverse. Treatments exist, but for advanced cancers, such as advanced laryngeal cancer, the 5-year survival rate is only around 40%. HNC also affects the face and throat, which can cause breathing problems, difficulty swallowing, voice changes, and significant impact on quality of life.

The effectiveness of treatment is limited by tumor diversity and complex interactions between cancer cells, immune cells, and surrounding tissue (tumor microenvironment, TME). Most research so far comes from Western populations, but genetic and viral differences in Asian patients require domestic studies. To provide personalized treatment, it is essential to collect clinical and genetic data from Korean patients and study their tumors and TME.

Need for Long-term Follow-up Studies Even early-stage HNC can recur locally, with recurrence rates reported between 20-57%. Recurrent or metastatic HNC has poor prognosis, with only 20-30% surviving five years. HNC usually progresses from pre-cancerous lesions to primary tumors and then spreads to lymph nodes. The molecular mechanisms behind this progression are not fully understood.

Various factors including smoking, alcohol, and HPV infection influence HNC development. HPV-positive patients show better outcomes, but their immune response may be suppressed. Therefore, continuous observation of HNC patients from early disease to recurrence is necessary to identify biomarkers that predict outcomes and to find more effective treatments.

Importance of Studying Tumor Microenvironment Immune checkpoint inhibitors (ICIs) combined with chemotherapy have improved survival in HNC. For example, pembrolizumab plus chemotherapy extended median overall survival to 13 months versus 10.7 months with standard treatment. Patients with higher PD-L1 expression responded better, but some high PD-L1 patients still did not respond, and some low PD-L1 patients responded well. Clear biomarkers to predict who will benefit from ICIs are still lacking.

Role of Samsung Medical Center In Korea, about 3,000 new cases of lip, oral, and throat cancer occur annually. Samsung Medical Center treated 550 of these patients in 2021, about one-fifth of national cases. More than half presented with advanced disease. Five-year survival rates for patients at Samsung Medical Center are higher than national averages: 78.5% overall, 93.2% for local tumors, and 37.8% for metastatic disease. These data show the importance of collecting patient information and samples for ongoing research.

Study Objectives

This study aims to:

Collect clinical information from HNC patients at Samsung Medical Center.

Collect tissue and blood samples at diagnosis, before and during treatment, and at disease progression or suspected recurrence.

Identify biomarkers that can guide personalized treatment in the future.

Study Design Eligibility

Inclusion Criteria:

Adults 20 years or older.

Histologically confirmed HNC at any head and neck site (oral cavity, pharynx, larynx, nasal cavity, salivary glands, or other locations). Patients diagnosed elsewhere are eligible if pathology is confirmed at Samsung Medical Center.

Various HNC-related cancer types including squamous cell carcinoma, adenocarcinoma, undifferentiated carcinoma, and others.

Scheduled for or previously received appropriate treatment (surgery, radiotherapy, chemotherapy, or immunotherapy).

Able to understand and sign informed consent.

Exclusion Criteria:

Not meeting inclusion criteria.

Any other reason deemed unsuitable by the investigator.

Sample Size:

Approximately 350 patients per year will participate, based on the number undergoing biopsy and blood collection at Samsung Medical Center.

Duration The study will last 60 months from IRB approval (~December 31, 2030).

Data and Sample Collection

Clinical Data:

Collect demographics, diagnosis details (location, stage, HPV status), medical history, smoking/alcoh

DETAILED DESCRIPTION:
1. Background and Rationale 1.1 Need for Personalized Precision Medicine in Head and Neck Cancer Head and neck cancer (HNC) ranks as the sixth leading cause of cancer-related death, with over 650,000 new cases diagnosed worldwide each year. Approximately 60% of HNC patients present with locally advanced disease at diagnosis, and many experience recurrence or metastasis despite multimodal therapy . Major risk factors include tobacco and alcohol use, prior radiation therapy, and infection with human papillomavirus (HPV).

   Prognostic differences across racial groups are partly explained by the prevalence of HPV-associated disease and genetic factors. HPV infection is commonly observed in oropharyngeal cancers, particularly tonsillar cancers. Patients with HPV-positive oropharyngeal cancer generally respond better to treatment and have improved overall survival compared to HPV-negative patients. Conversely, epidermal growth factor receptor (EGFR) amplification is associated with poorer prognosis.

   HNC arises in diverse anatomical sites, including the oral cavity, pharynx, larynx, nasal cavity, nasopharynx, and salivary glands. Although squamous cell carcinoma is the most common subtype due to tobacco exposure, other histologies such as salivary gland carcinoma, adenoid cystic carcinoma, and others contribute to clinical heterogeneity.

   Although multimodal treatment-including surgery, radiation, and chemotherapy-is currently applied, outcomes for advanced laryngeal cancer remain limited, with 5-year overall survival (OS) around 40%. Moreover, HNC often affects the face and laryngeal region, significantly impairing quality of life by causing disfigurement, breathing difficulties, dysphagia, and voice disorders.

   Therapeutic efficacy is further limited by intra- and inter-tumoral heterogeneity and complex interactions within the tumor microenvironment (TME). Existing HNC research primarily reflects Western populations, whereas differences in subtype distribution, etiology, viral prevalence, and genetics in Asian populations necessitate localized data collection. Therefore, molecular and genetic analyses of domestic patient samples, along with TME research, are essential to implement personalized precision medicine in HNC.

   1.2 Need for Longitudinal Follow-up Studies in Head and Neck Cancer Major causes of death in patients with advanced HNC include local recurrence, cervical lymph node metastasis, and resistance to systemic therapy. Even early-stage HNC has a reported local recurrence rate of 20-57%, and despite adjuvant chemoradiotherapy, the 5-year local recurrence rate remains approximately 30%. Recurrent or metastatic HNC carries a poor prognosis, with 5-year survival rates of only 20-30%.

   For squamous cell carcinoma of the head and neck (HNSCC), disease progression typically follows a stepwise sequence from precancerous leukoplakia in normal tissue, to primary carcinoma, and ultimately to lymph node metastasis. While studies have sought to identify markers predicting malignant transformation, molecular mechanisms remain unclear.

   HNSCC pathogenesis is multifactorial, involving tobacco, alcohol, and HPV infection. HPV is particularly influential in disease progression, and HPV-positive oropharyngeal cancer patients generally exhibit favorable outcomes. Genetic studies indicate that both innate and adaptive antiviral immune responses are suppressed in HPV-positive patients.

   Thus, continuous monitoring of clinical progression and tumor characteristics from early-stage disease to local recurrence or metastasis is critical to identify prognostic biomarkers and guide effective therapies.

   1.3 Need for Tumor Microenvironment Research in Head and Neck Cancer Combination therapy with immune checkpoint inhibitors (ICIs) and chemotherapy has significantly improved overall survival. In the KEYNOTE-048 study, patients receiving pembrolizumab plus platinum-based chemotherapy achieved a median OS of 13.0 months, compared to 10.7 months for cetuximab plus chemotherapy (HR 0.71, 95% CI 0.59-0.85) over a median follow-up of 45 months. In patients with PD-L1 combined positive score (CPS) ≥20, HR was 0.62 (95% CI 0.46-0.84), and for CPS ≥1, HR was 0.64 (95% CI 0.53-0.78). Subgroup analysis showed that PD-L1 CPS correlated with OS in the pembrolizumab group, but not in the cetuximab group.

   Despite the introduction of ICIs, only 15-26% of patients respond well. Some patients with high PD-L1 do not respond, while a subset of low PD-L1 patients shows prolonged response. Biomarkers predicting ICI responders remain unclear.

   1.4 Role of Samsung Medical Center in Head and Neck Cancer Research According to the 2021 cancer registry, approximately 3,000 cases of lip, oral cavity, and pharyngeal cancers were reported in Korea. In the same year, Samsung Medical Center recorded 550 cases, representing about one-fifth of national cases. The number of HNC cases at Samsung Medical Center continues to increase, with over half presenting as locally advanced disease. The 5-year survival rate for these patients is 78.5%, with localized tumors achieving 93.2% and distant metastases 37.8%. This is superior to national outcomes, highlighting the need for longitudinal follow-up and research using Samsung Medical Center patient data.

   ________________________________________
2. Study Objectives

The study aims to:

1. Collect clinical information from HNC patients visiting Samsung Medical Center.
2. Prospectively collect tissue and blood samples at initial diagnosis, before and during treatment, at disease progression, and upon suspected recurrence.
3. Identify biomarkers to support future personalized medicine approaches. ________________________________________

3. Study Design 3.1 Eligibility Criteria Inclusion Criteria

1. Age ≥20 years.
2. Histologically confirmed head and neck cancer, including tumors of the oral cavity, pharynx, larynx, nasal cavity, salivary glands, and other HNC sites. Patients diagnosed elsewhere are eligible if pathology is confirmed at Samsung Medical Center.
3. Histologic types include squamous cell carcinoma, undifferentiated carcinoma, poorly differentiated carcinoma, non-keratinizing carcinoma, adenocarcinoma, carcinoma of unknown primary in HNC, salivary gland cancer, malignant melanoma or sarcoma of the head and neck, and other relevant malignancies.
4. Patients scheduled for or having received appropriate HNC treatment (surgery, radiotherapy, cytotoxic chemotherapy, or immune checkpoint inhibitors).
5. Written informed consent obtained. Exclusion Criteria

1. Failure to meet inclusion criteria. 2. Other reasons deemed by the investigator to make the patient unsuitable for study participation.

Target Sample Size Approximately 350 patients per year are expected to undergo biopsy and blood sampling at Samsung Medical Center.

________________________________________ 3.2 Study Duration 60 months from IRB approval (~December 31, 2030).

________________________________________ 3.3 Study Procedures 3.3.1 Data Collection Clinical data and questionnaires will be collected from patients who provide informed consent. Tissue and blood samples will be collected prospectively at baseline, during treatment, at disease progression, and upon recurrence.

1. Clinical Data: Demographics, diagnosis (date, site, pathology, stage, HPV/P16 status), medical history, smoking/alcohol history, treatment details (surgery, radiation, chemotherapy), treatment response, progression, and survival will be collected. For patients not attending follow-up visits, survival and treatment information will be obtained via phone.
2. Tissue Collection: Fresh tissue will be collected when possible. Residual diagnostic or therapeutic samples stored in pathology may be used. During follow-up, tissue obtained for suspected recurrence will be stored, along with samples collected for treatment response assessment. Normal tissue distant from tumor, adjacent normal tissue, tumor tissue, and lymph nodes will be collected during surgery.
3. Blood Collection: Blood samples will be collected before treatment, during follow-up, at disease progression, and at imaging assessments. For patients receiving concurrent chemoradiotherapy (CCRT), blood will be collected before treatment, 3 weeks post-treatment (±1 week), 6 weeks post-treatment (±1 week), during imaging follow-up, and at progression. For patients receiving immune checkpoint inhibitors, blood will be collected at baseline, 3 weeks (±1), 6 weeks (±1), 12 weeks (±3), and at subsequent imaging assessments, with 20-30 mL per collection. Samples will be stored in secure, designated freezers.
4. Questionnaires: Administered at baseline, post-treatment, 3 months post-treatment, and every 6 months for 5 years. Items include demographics, lifestyle, medical history, pain, psychological status, quality of life (EORTC C30+HN35), PHQ-9, and social support.

3.3.2 Laboratory Analysis

* Tissue: WGS and WTS to characterize tumors; single-cell sequencing, spatial transcriptomics, or multiplex immunofluorescence for TME analysis. Immune cell populations (T cells, B cells, neutrophils, macrophages), immune gene signatures (IFN, IL family), T-cell subsets (CD4+, CD7+, CD8+, CD16, CD34+, CD38+, D56+), and PD-1/PD-L1 expression will be assessed pre- and post-treatment.
* Blood: WGS as normal reference, WTS for immune cell profiling, and ctDNA analysis for minimal residual disease (MRD).

3.3.3 Sample Management Samples will be stored with coded identifiers. De-identified samples may be sent to external laboratories; access to identifiers will be limited. Samples will be retained for 20 years or according to participant-specified duration. Post-study, external samples will be returned or destroyed. Samples with irreversibly anonymized identifiers will be handled per applicable regulations.

3.3.4 Future Research Use

* Sample Management: With participant consent, leftover samples may be stored for exploratory research without additional collection. External research may be performed by investigators not part of this study, using coded samples, which will be returned or destroyed after analysis.
* Data Management: With participant consent, de-identified clinical and genomic data (WES, WTS, WGS raw and analyzed data) may be used for future exploratory research. External institutions may receive coded data for analysis; identifiers will remain inaccessible.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 years or older

  * Histologically confirmed head and neck cancer (including cancers of the oral cavity, pharynx, larynx, nasal cavity, salivary glands, and other head and neck sites) Patients diagnosed at outside institutions but pathologically confirmed as head and neck cancer at Samsung Medical Center are also eligible.)

    * Patients with similar histologic types (including squamous cell carcinoma, undifferentiated carcinoma, poorly differentiated carcinoma, nonkeratinizing carcinoma, and adenocarcinoma), as well as cancers of unknown primary, salivary gland cancers, head and neck malignant melanoma, sarcomas, and other malignancies are eligible.

      * Diagnosed with head and neckk cancer and scheduled to receive, or previously received, appropriate treatment (radiation therapy, cytotoxic chemotherapy, immune checkpoint inhibitors, or surgery).

        * Ability to understand the purpose of the study and willingness to sign informed consent.

Exclusion Criteria:

* Any other condition that, in the opinion of the investigator, makes the patient unsuitable for study participation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 550 head and neck cancer patients visit Samsung Medical Center annually, and approximately 350 patients seek biopsy and other tests in a capable, primary care setting. Therefore, we plan to conduct this study on approximately 350 medical professionals annually.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival(OS) | From study enrollment until death from any cause, assessed up to study completion (approximately 5 years.)
  Overall survival is defined as the time from the date of study enrollment to the date of death from any cause. Survival will be analyzed using Kaplan-Meier survival plots, and the effect of clinical and treatment-realated variables on survival will be assessed using Cox's proportional hazard model and Log-rank test. A p-value <0.05 will be considered statistivally significant.

SECONDARY OUTCOMES:
Disease-Free Survival(DFS) | From treatment completion until disease recurrence or death from any cause, assessed up to study completion (approximately 5 years).
  DFS is defined as the time from treatment completion to the first documented recurrence or death. Kaplan-Meier plots and Cox's proportional hazard model will be used for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Privacy and Security IPD information represents an individual's characteristics, so sharing it may pose a risk of personal information leakage.

REFERENCES:
- [Background] Kumar B, Cordell KG, Lee JS, Worden FP, Prince ME, Tran HH, Wolf GT, Urba SG, Chepeha DB, Teknos TN, Eisbruch A, Tsien CI, Taylor JM, D'Silva NJ, Yang K, Kurnit DM, Bauer JA, Bradford CR, Carey TE. EGFR, p16, HPV Titer, Bcl-xL and p53, sex, and smoking as indicators of response to therapy and survival in oropharyngeal cancer. J Clin Oncol. 2008 Jul 1;26(19):3128-37. doi: 10.1200/JCO.2007.12.7662. Epub 2008 May 12. PMID 18474878
- [Background] Vermorken JB, Remenar E, van Herpen C, Gorlia T, Mesia R, Degardin M, Stewart JS, Jelic S, Betka J, Preiss JH, van den Weyngaert D, Awada A, Cupissol D, Kienzer HR, Rey A, Desaunois I, Bernier J, Lefebvre JL; EORTC 24971/TAX 323 Study Group. Cisplatin, fluorouracil, and docetaxel in unresectable head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1695-704. doi: 10.1056/NEJMoa071028. PMID 17960012
- [Background] Seiwert TY, Salama JK, Vokes EE. The concurrent chemoradiation paradigm--general principles. Nat Clin Pract Oncol. 2007 Feb;4(2):86-100. doi: 10.1038/ncponc0714. PMID 17259930
- [Background] Seiwert TY, Salama JK, Vokes EE. The chemoradiation paradigm in head and neck cancer. Nat Clin Pract Oncol. 2007 Mar;4(3):156-71. doi: 10.1038/ncponc0750. PMID 17327856
- [Background] Posner MR, Hershock DM, Blajman CR, Mickiewicz E, Winquist E, Gorbounova V, Tjulandin S, Shin DM, Cullen K, Ervin TJ, Murphy BA, Raez LE, Cohen RB, Spaulding M, Tishler RB, Roth B, Viroglio Rdel C, Venkatesan V, Romanov I, Agarwala S, Harter KW, Dugan M, Cmelak A, Markoe AM, Read PW, Steinbrenner L, Colevas AD, Norris CM Jr, Haddad RI; TAX 324 Study Group. Cisplatin and fluorouracil alone or with docetaxel in head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1705-15. doi: 10.1056/NEJMoa070956. PMID 17960013
- [Background] Bonner JA, Harari PM, Giralt J, Azarnia N, Shin DM, Cohen RB, Jones CU, Sur R, Raben D, Jassem J, Ove R, Kies MS, Baselga J, Youssoufian H, Amellal N, Rowinsky EK, Ang KK. Radiotherapy plus cetuximab for squamous-cell carcinoma of the head and neck. N Engl J Med. 2006 Feb 9;354(6):567-78. doi: 10.1056/NEJMoa053422. PMID 16467544
- [Background] Leemans CR, Braakhuis BJ, Brakenhoff RH. The molecular biology of head and neck cancer. Nat Rev Cancer. 2011 Jan;11(1):9-22. doi: 10.1038/nrc2982. Epub 2010 Dec 16. PMID 21160525
- See also: Hah, J. H. (2012). Personalized Treatment of Head and Neck Cancers and the Role of Head and Neck Surgeons. Korean Journal of Otorhinolaryngology-Head and Neck Surgery, 55(8), 471-475. — https://www.koreamed.org/SearchBasic.php?RID=2277369